CLINICAL TRIAL: NCT04155372
Title: Effect of Different Fluid Ingestion Rate on Post-exercise Rehydration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, LIN, JIAN-YU, Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS19-CT7-08
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Dehydration
Keywords: sports nutrition; dehydration; sports medicine; rehydration; ingestion rate
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30min (Experimental): The participants arrived to the trials euhydrated and were dehydrated to 2% of body weight (BW) by running. After a rest, they ingested sports drink in a volume equivalent to 150% of BW loss in 30 min.
  Interventions: Procedure: Different Fluid Ingestion Rate
- 60min (Experimental): The participants arrived to the trials euhydrated and were dehydrated to 2% of body weight (BW) by running. After a rest, they ingested sports drink in a volume equivalent to 150% of BW loss in 60 min.
  Interventions: Procedure: Different Fluid Ingestion Rate
- 90min (Experimental): The participants arrived to the trials euhydrated and were dehydrated to 2% of body weight (BW) by running. After a rest, they ingested sports drink in a volume equivalent to 150% of BW loss in 90 min.
  Interventions: Procedure: Different Fluid Ingestion Rate

INTERVENTIONS:
Procedure: Different Fluid Ingestion Rate — The participants ingested sports drink in a volume equivalent to 150% of BW loss, in 30 min, 60 min, or 90min.

SUMMARY:
The purpose of the present study is to investigate the effect of different rate of fluid consumption on post-exercise rehydration.

DETAILED DESCRIPTION:
The body water deficits equivalent to 2% body mass might impair performance. Due to high exercise intensity, thermal environment, or rule limitation, athletes often in dehydration status post-exercise. Thus, how to rehydrate effectively to prepare the next game is important. The participants arrived to the lab euhydrated and were dehydrated to 2% of body weight by running. After a rest, they will ingest sports drink in a volume equivalent to 150% of BW loss in 30 min, 60 min, or 90 min. Urine and blood sample will be collected to evaluate hydration status.

ELIGIBILITY:
Inclusion Criteria:

* 20~35 years old male
* Exercise 150 min per week
* Without chronic disease or gastrointestinal surgery

Exclusion Criteria:

* Injury
* Answer "Yes" in part 1 of the Physical Activity Readiness Questionnaire(PAR-Q+)
* Participate in other studies within one month

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
specific gravity of urine(SG) | Change from baseline outcome measure at dehydration and 1st and 2nd hour in recovery period
  dehydration: >= 1.020
Osmolality(Urine) | Change from baseline outcome measure at dehydration and 1st and 2nd hour in recovery period
  dehydration: >= 700 mosm/kg
Osmolality(Blood) | Change from baseline outcome measure at dehydration and 1st and 2nd hour in recovery period
  dehydration: >= 290 mosm/kg
Vasopressin | Change from baseline outcome measure at dehydration and 1st and 2nd hour in recovery period
  Vasopressin, also called antidiuretic hormone (ADH), arginine vasopressin (AVP) or argipressin, is a hormone synthesized as a peptide prohormone in neurons in the hypothalamus, and is converted to AVP. Increasing the water reabsorption and excretion of more concentrated urine.
sodium(blood) | Change from baseline outcome measure at dehydration and 1st and 2nd hour in recovery period
  135~145mEq/L
Body weight change | Change from baseline outcome measure at dehydration and 1st and 2nd hour in recovery period
  measure body weight at baseline, dehydration, 1st and 2nd hour in recovery period in kg

CONTACTS AND LOCATIONS:
Overall Officials: JIAN-YU LIN, Principal Investigator — Kaohsiung Veterans General Hospital.